CLINICAL TRIAL: NCT02299856
Title: Cardiac Magnetic Resonance in Acute Myocarditis
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Claas P. Naehle, PD Dr. med., University Hospital, Bonn
Other Study IDs: 150/13.2
Record Dates: First submitted 2014-11-13; First posted 2014-11-24 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Myocarditis
Keywords: Magnetic Resonance Imaging; Diagnostic Imaging
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hematocrit is obtained prior to cardiac MR.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Myocarditis: Patients with strong clinical evidence for acute myocarditis (recent infection, elevated troponin and white blood cell count).
  Interventions: Other: Cardiac magnetic resonance scan
- Healthy Controls: Healthy volunteers without any signs of cardiac disease.
  Interventions: Other: Cardiac magnetic resonance scan

INTERVENTIONS:
Other: Cardiac magnetic resonance scan

SUMMARY:
Cardiac magnetic resonance (MR) is an established noninvasive diagnostic tool for detection of acute myocarditis. Diagnosis of myocarditis at 1.5T is currently made with the help of the Lake Louise Criteria (two of three criteria have to be positive in order to establish the diagnosis). Although these criteria are accepted and widely used in clinical routine, several disadvantages exist. Newer parameters like myocardial T1 and T2 mapping, extracellular volume fraction (ECV) and myocardial strain analysis have the potential to complement or even replace some of the Lake Louise Criteria and further enhance the diagnostic performance of cardiac MR in patients suspected of having acute myocarditis. The aim of our study is to evaluate the diagnostic performance of a comprehensive cardiac MR protocol in patients with acute myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* No past medical history of cardiac disease.
* No cardiovascular risk factors (e.g. diabetes or hypertension)

Exclusion Criteria:

* Contraindications for cardiac MR

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients are included in the myocarditis group if they showed clinical evidence of acute myocarditis(acute chest pain, history of viral infection, elevated white blood cell count, ECG changes and/or elevated troponin).
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Myocardial T1 relaxation time | Measurement will be performed within 2 weeks after MRI scan.
  Changes in myocardial T1 relaxation time is of interest in patients with acute myocarditis. T1 relaxation times will be directly obtained from the T1 maps through ROI analysis. T1 maps will be analyzed using a segmental approach. T1 relaxation times are given in [ms].
Myocardial T2 relaxation time | Measurement will be performed within 2 weeks after MRI scan.
  Changes in myocardial T2 relaxation time is of interest in patients with acute myocarditis. T2 relaxation times will be directly obtained from T2 maps through ROI analysis. T2 maps will be analyzed using a segmental approach. T2 relaxation times are given in [ms].
Myocardial ECV measurements | Measurement will be performed within 2 weeks after MRI scan.
  Changes in myocardial ECV parameters is of interest in patients with acute myocarditis. Hematocrit corrected ECV will be calculated using pre- and post-contrast T1 values for myocardium and blood pool using following formula:
  ECV= (1⁄T1 "myocardium post contrast"-1⁄T1 "myocadium pre contrast")/(1⁄T1 "blood post contrast"-1⁄ T1 "blood pre contrast") x (1-hematocrit).
  ECV is given in percentage.
Myocardial strain analysis (focussed on longitudinal strain) | Measurement will be performed within 2 weeks after MRI scan.
  Changes in longitudinal strain as determined by echocardiography has been described in patient with acute myocarditis. In our study longitudinal strain is measured using feature tracking, which allows for strain calculation from standard MR cine datasets.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn, Dept. of Radiology, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Luetkens JA, Doerner J, Thomas DK, Dabir D, Gieseke J, Sprinkart AM, Fimmers R, Stehning C, Homsi R, Schwab JO, Schild H, Naehle CP. Acute myocarditis: multiparametric cardiac MR imaging. Radiology. 2014 Nov;273(2):383-92. doi: 10.1148/radiol.14132540. Epub 2014 Jun 6. PMID 24910904
- [Derived] Luetkens JA, Homsi R, Sprinkart AM, Doerner J, Dabir D, Kuetting DL, Block W, Andrie R, Stehning C, Fimmers R, Gieseke J, Thomas DK, Schild HH, Naehle CP. Incremental value of quantitative CMR including parametric mapping for the diagnosis of acute myocarditis. Eur Heart J Cardiovasc Imaging. 2016 Feb;17(2):154-61. doi: 10.1093/ehjci/jev246. Epub 2015 Oct 16. PMID 26476398